CLINICAL TRIAL: NCT06968663
Title: Electrical Field Guided Transcranial Magnetic Stimulation to Treat Subacute Post-stroke Aphasia
Brief Title: Transcranial Magnetic Stimulation + Language Therapy to Treat Subacute Aphasia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 856766
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Stroke; Aphasia; Aphasia Following Cerebral Infarction
Keywords: aphasia; stroke; Transcranial Magnetic Stimulation; Non-invasive brain stimulation; language therapy
MeSH Terms: conditions — Stroke; Aphasia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real TMS (Experimental): Some of our participants will be randomized to the real treatment arm where they will receive 10 sessions of real TMS paired with language therapy.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS); Behavioral: Modified Constraint Induced Language Therapy (mCILT)
- Fake TMS (Sham Comparator): Some of our participants will be randomized to the sham treatment arm where they will receive 10 sessions of fake TMS paired with language therapy.
  Interventions: Behavioral: Modified Constraint Induced Language Therapy (mCILT)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — TMS, is a form of non-invasive brain stimulation, that uses magnetic pulses to stimulate specific areas of the brain. In this study we will utilize theta-burst stimulation which uses a higher frequency pulse of 50 Hz delivered for 40 seconds for a total of 600 pulses.
  Arms: Real TMS
Behavioral: Modified Constraint Induced Language Therapy (mCILT) — Constraint-induced language therapy (CILT) is a treatment approach for aphasia that focuses on forcing the patient to use their impaired language skills, while restricting the use of compensatory strategies like gestures or writing. All participants will receive mCILT.

SUMMARY:
The goal of this clinical trial is to determine if Transcranial Magnetic Stimulation (TMS) combined with modified Constraint Induced Language Therapy (mCILT) is an effective treatment for aphasia when delivered in the subacute stage after stroke.

The main questions this study aims to answer are:

1. Can TMS combined with mCILT improve overall speech?
2. Can we identify specific behavioral and biological characteristics that would benefit most from the TMS and mCILT treatment?

Researchers will compare real TMS to sham (fake) TMS to see whether TMS can treat subacute aphasia.

Importantly, this trial will use electric field guided TMS to identify optimal and individualized stimulation intensity and site targeting.

Participants will:

* Complete a screening and medical intake to determine eligibility
* Undergo MRI scans
* Participate in 10 consecutive sessions (Monday-Friday) of TMS and mCILT treatment
* Complete follow-up assessments immediately and 4 months after treatment

DETAILED DESCRIPTION:
Aphasia is an acquired disorder of language that occurs in approximately 30% of individuals with stroke and impacts approximately 1 million Americans (see NINDS.NIH.gov). Current treatments for aphasia are only modestly beneficial, so there is a clear need for more efficacious therapy.

Most studies of TMS as a therapy for aphasia have investigated treatment in the chronic phase after stroke (>6 months post-stroke). Previous research has demonstrated that TMS improves language performance in persons with chronic aphasia and the benefit has been shown to be sustained. Several lines of evidence, however, suggest that TMS treatment in the subacute period may be more effective than interventions in the chronic stage.

One limitation of TMS has been variability in response; TMS has shown good within-subject reliability but more substantial variability between subjects. In recognition of these issues, "electrical field" (e-field) models have been developed to account for these individual differences in anatomy. We will the utilize e-field models in conjunction with an individually determined resting motor threshold to generate a personalized treatment regimen that is likely to ensure that all subjects receive the same TMS intensity relative to their individual motor threshold and greatly reduces the possibility of under- or over-dosing with respect to TMS intensity. We will employ continuous theta-burst stimulation, 600 brief electrical pulses delivered in 40 seconds, over the right front part of the brain (pars triangularis).

Participants who are enrolled can expect to undergo a battery of tests to define their language function as well as a research MRI scan that will be used to guide TMS therapy and to assess the size and location of the stroke and its impact on brain pathways. After baseline testing, subjects will undergo treatment using TMS (or sham) + mCILT for 10 sessions (Monday-Friday) over the course of 2 consecutives week. Follow-up assessment of language functioning will be assessed immediately and 4 months after treatment.

Participants will be compensated for their time and travel.

ELIGIBILITY:
Inclusion Criteria:

* Left hemisphere stroke resulting in aphasia
* The stroke must have occurred between 2 and 6 weeks prior to enrollment
* Must be able to understand the nature of the study, and give informed consent
* English proficiency
* Right-handed

Exclusion Criteria:

* History of serious and/or ongoing issues with substance abuse
* Previous head trauma with loss of consciousness for more than 5 minutes
* History of major psychiatric illness
* Dementia, or other neurological conditions
* Epilepsy, or seizure after the stroke event
* Pacemaker
* Diagnosis of tinnitus
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Overall language function | From Baseline to 4 months post-interventions
  Change in performance on the Western Aphasia Battery (WAB-AQ score). WAB AQ Score is out of 100, where a higher score means less language impairment.

CONTACTS AND LOCATIONS:
Overall Officials: H. Branch Coslett, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
No, the study team does not plan to share participating data at this time.